CLINICAL TRIAL: NCT01462500
Title: Pharmacokinetics of Miltefosine in Children and Adults: Implications for the Treatment of Cutaneous Leishmaniasis in Colombia.
Brief Title: Pharmacokinetics of Miltefosine in Children and Adults
Acronym: PK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Internacional de Entrenamiento e Investigaciones Médicas (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2229-519-28930
Record Dates: First submitted 2011-10-25; First posted 2011-10-31 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Miltefosine; pharmacokinetics; cutaneous leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — miltefosine; Pharmacogenomic Variants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Miltefosine (Experimental): Miltefosine PO at a dose of 1.8-2.5 mg/kg/day for 28 days
  Interventions: Drug: Miltefosine

INTERVENTIONS:
Drug: Miltefosine — Children (2-12 years of age) and adults (18-60 years of age) will receive Miltefosine PO at a dose of 1.8-2.5 mg/kg/day for 28 days.
  Other Names: pharmacokinetic

SUMMARY:
The purpose of this study is to determine the pharmacokinetics of miltefosine in children and adults with cutaneous leishmaniasis in plasma and intracellularly, and its relation with the parasitologic response. The results will provide pharmacologic bases to optimize the use of miltefosine for the treatment of cutaneous leishmaniasis, and will provide the knowledge base to assess the impact of pharmacokinetic behavior in children and adults on the emergence of drug resistance.

DETAILED DESCRIPTION:
An open-label phase IV clinical trial of miltefosine, designed to evaluate intracellular and plasma drug pharmacokinetics in children and adults using a population pharmacokinetics design. Two study groups have been defined: 1) children 2-12 years of age (n=30) and 2) adults 18-60 years of age (n=30) with confirmed parasitological diagnosis of cutaneous leishmaniasis. The participants will receive supervised standard treatment with miltefosine: 1.8 - 2.5 mg/Kg of weight for 28 days.

Miltefosine concentration will be determined in plasma and Peripheral Blood Mononuclear Cell (PBMCs), from 3 or 10ml peripheral blood samples in children and adults respectively. Sampling will be conducted pre-dosing at days 0,1,15 and 29 during treatment, and at months 1, 2, 3 and 6 post-treatment.

A population pharmacokinetics analysis will be performed using a non-linear model of mixed effects with the software Nonlinear Mixed-effects Model (NONMEM), R and Piranha. Parasite burden will be determined by 7SLRNA Quantitative Polymerase Chain Reaction (qPCR) of Leishmania from swab samples of lesions and extralesional tissues before and at the end of treatment. The relationship between pharmacokinetics and parasite persistence/burden will be determined by correlation analysis and pharmacodynamic modeling.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2-12 years of age, or 18-60 years of age
* Weight greater than 10 kg
* Parasitologic confirmation of cutaneous leishmaniasis
* Normal hepatic and kidney function

Exclusion Criteria:

* Pregnant or lactating women, and women who are planning to conceive during the study or that reject the use of birth control methods.
* Use of drugs with antileishmanial potential during the previous 6 months, including pentavalent antimonials, amphotericin B, miltefosine, and pentamidine
* Mucocutaneous or visceral leishmaniasis
* For female children, menses or other evidence of reproductive maturity

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Intracellular and plasma concentration of miltefosine | Participants will be followed up to 26 weeks.
Parasite burden in lesions and extralesional tissues. | Participants will be followed up to 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nancy C Saravia, PhD, Principal Investigator — Centro Internacional de Entrenamiento e Investigaciones Médicas, CIDEIM
Locations (1):
- Corporación Centro Internacional de entrenamiento e Investigaciónes Médicas, Cali, Valle del Cauca Department, Colombia

REFERENCES:
- [Background] Sindermann H, Engel J. Development of miltefosine as an oral treatment for leishmaniasis. Trans R Soc Trop Med Hyg. 2006 Dec;100 Suppl 1:S17-20. doi: 10.1016/j.trstmh.2006.02.010. Epub 2006 May 26. PMID 16730362
- [Background] Dorlo TP, van Thiel PP, Huitema AD, Keizer RJ, de Vries HJ, Beijnen JH, de Vries PJ. Pharmacokinetics of miltefosine in Old World cutaneous leishmaniasis patients. Antimicrob Agents Chemother. 2008 Aug;52(8):2855-60. doi: 10.1128/AAC.00014-08. Epub 2008 Jun 2. PMID 18519729
- [Background] Anderson BJ, Allegaert K, Holford NH. Population clinical pharmacology of children: general principles. Eur J Pediatr. 2006 Nov;165(11):741-6. doi: 10.1007/s00431-006-0188-y. Epub 2006 Jun 29. PMID 16807730
- [Background] Berman JJ. Treatment of leishmaniasis with miltefosine: 2008 status. Expert Opin Drug Metab Toxicol. 2008 Sep;4(9):1209-16. doi: 10.1517/17425255.4.9.1209. PMID 18721114
- [Derived] Castro MDM, Cossio A, Velasco C, Osorio L. Risk factors for therapeutic failure to meglumine antimoniate and miltefosine in adults and children with cutaneous leishmaniasis in Colombia: A cohort study. PLoS Negl Trop Dis. 2017 Apr 5;11(4):e0005515. doi: 10.1371/journal.pntd.0005515. eCollection 2017 Apr. PMID 28379954
- [Derived] Castro MD, Gomez MA, Kip AE, Cossio A, Ortiz E, Navas A, Dorlo TP, Saravia NG. Pharmacokinetics of Miltefosine in Children and Adults with Cutaneous Leishmaniasis. Antimicrob Agents Chemother. 2017 Feb 23;61(3):e02198-16. doi: 10.1128/AAC.02198-16. Print 2017 Mar. PMID 27956421